CLINICAL TRIAL: NCT03021980
Title: Development and Evaluation of SuperFIT: Systems of Underprivileged Preschoolers in Their Home and Preschool EnviRonment: Family Intervention Trial.
Brief Title: Systems of Underprivileged Preschoolers in Their Home and Preschool EnviRonment: Family Intervention Trial
Acronym: SuperFIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Fonds NutsOhra (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NL58061.068.16
Record Dates: First submitted 2017-01-09; First posted 2017-01-16 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-03

CONDITIONS: Child Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — 3-methylfentanyl isothiocyanate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SuperFIT (Experimental): This is the intervention group. They will receive the intervention SuperFIT.
  Interventions: Behavioral: SuperFIT
- Control (No Intervention): This is the control group. Participants will receive 'care as usual' in this arm.

INTERVENTIONS:
Behavioral: SuperFIT — Behavioural intervention with two components. One component will consist of social and physical environmental changes at the preschools and the other component consists of a family educational program.
  Arms: SuperFIT

SUMMARY:
This study will evaluate the effectiveness of SuperFIT, an integrative lifestyle intervention for preschool children. It will consist of both an preschool component and a family component and is aimed at increasing healthy nutrition and physical activity. Half of the participating preschools will implement SuperFIT, while the other half of the preschools will continue as usual.

ELIGIBILITY:
Inclusion Criteria:

* children attending the participating preschools
* at least one parent has to be able to understand the Dutch language
* Both caregivers (if applicable) of the child give informed consent

Exclusion Criteria:

* There are no exclusion criteria for this study

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2017-01; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change in BMI | from baseline to one year and 1.5 years after baseline
Change in physical activity by an Actigraph accelerometer | from baseline to one year and 1.5 years after baseline
Change in Diet, Food and Nutrition by a 24HR recall | from baseline to one year and 1.5 years after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sanne Gerards, Dr., Principal Investigator — Department of Health Promotion, Maastricht University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van de Kolk I, Gerards S, Verhees A, Kremers S, Gubbels J. Changing the preschool setting to promote healthy energy balance-related behaviours of preschoolers: a qualitative and quantitative process evaluation of the SuperFIT approach. Implement Sci. 2021 Dec 4;16(1):101. doi: 10.1186/s13012-021-01161-9. PMID 34863245